CLINICAL TRIAL: NCT01703247
Title: Ganglionated Plexi Ablation vs Linear Ablation in Patients Undergoing Pulmonary Vein Isolation for Persistent/Longstanding Persistent Atrial Fibrillation: A Randomized Comparison
Brief Title: Ganglionated Plexi Ablation Combined With Pulmonary Vein Isolation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GP-LL-AF
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Arrhythmias; Ablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVI+LL (Active Comparator): Circumferential PVI was accomplished and then additional ablation lines were created by connecting the left inferior PV to the mitral annulus (mitral isthmus) and the LA between the two superior PVs (roof). Finally, patients underwent cavo-tricuspid isthmus ablation in the right atrium.
  Interventions: Procedure: Pulmonary vein isolation; Procedure: Linear Lesion Ablation
- PVI+GP (Active Comparator): To accomplish ganglionated plexi ablation, LA target sites were identified as the anatomic locations where vagal reflexes were evoked by transcatheter high-frequency stimulation (HFS). Rectangular electrical stimuli were delivered at a frequency of 20-50 Hz, output amplitude 15 V and pulse duration of 10 ms, for 5 sec (Stimulator B-53, Biotok Inc, Russia).
  Interventions: Procedure: Pulmonary vein isolation; Procedure: Ganglionated plexi ablation

INTERVENTIONS:
Procedure: Pulmonary vein isolation
Procedure: Ganglionated plexi ablation
  Arms: PVI+GP
Procedure: Linear Lesion Ablation
  Arms: PVI+LL

SUMMARY:
The investigators have conducted a prospective, double-blind, randomized study to assess the comparative safety and efficacy of two different ablation strategies, PVI plus linear lesions (LL) versus PVI plus GP ablation, in patients with persistent or longstanding persistent AF. Results were assessed after follow-up of at least 3 years with the use of an implanted monitoring device (IMD).

ELIGIBILITY:
Inclusion Criteria:

* Persistent and longstanding persistent AF

Exclusion Criteria:

* congestive heart failure
* LV ejection fraction < 35%
* left atrial diameter > 60 mm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
freedom of atrial tachyarrhythmia, including AF and atrial flutter/tachycardia | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of CIrculation Pathology, Novosibirsk, Russia

REFERENCES:
- See also: State Research Institute of Circulation Pathology Official Site — http://www.meshalkin.ru/